CLINICAL TRIAL: NCT01949597
Title: Recurrences After Surgery for Deep Endometriosis Depending on the Involvement of the Surgical Margins in the Specimen
Status: Withdrawn | Type: Observational
Why Stopped: IP change Hospital
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Ignacio Rodriguez MSc, Epidemiologist, Fundacion Dexeus
Other Study IDs: DEX2013002
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2016-04

CONDITIONS: Deep Endometriosis; Recurrences; Margins in the Specimen; Laparoscopy; Prognosis Factors
MeSH Terms: conditions — Recurrence | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with symptomatic endometriosis
  Interventions: Procedure: laparoscopic surgery for deep endometriosis

INTERVENTIONS:
Procedure: laparoscopic surgery for deep endometriosis

SUMMARY:
The recurrence of endometriosis after surgery a formidable challenge for the gynecologist. Recurrence rates reported in the literature are very high, being 21.5% at 2 years and 40-50% at 5 years. Several theories attempt to explain these high figures. The three most widely accepted are:

* The presence of residual endometriotic tissue or residual endometriotic cells not completely eradicated during surgery
* The growth of undetected microscopic endometriosis during surgery
* The development of endometriotic lesions de novo Patients with symptomatic endometriosis diagnosed by ultrasound or MRI and suitable for surgery will participate in the study. The surgical specimens sent for pathology from bladder, vagina, uterosacral, sigma or rectum will be properly marked for studying the presence of endometriosis.

DETAILED DESCRIPTION:
Patients of Dexeus Universitary Institute that are having a laparoscopic surgery for deep endometriosis will participate in the study. A patient information sheet will be provided and written consent will be obtained. Patients who give written consent will participate in the trial. All patient information will be confidential and only be available to researches involved in the study.

Only three expert surgeons of the Gynecological Department of Dexeus Universitary Institute will participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptomatic endometriosis superior to 6 in a visual scale (VAS; Huskisson, 1974)diagnosed by ultrasound or MRI and suitable for laparoscopic surgery

Exclusion Criteria:

* previous surgeries for deep endometriosis
* Non complete surgery

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women with symptomatic deep endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-04 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Recurrences | Two years after surgery
  Evaluate clinical recurrence rate of endometriosis after complete surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Vazquez, MD, Principal Investigator — Hospital Quiron Dexeus
Locations (1):
- Departamento de Obstetricia Ginecologia y Reproducción. Institut Universitari Dexeus, Barcelona, Spain

REFERENCES:
- [Background] Guo SW. Recurrence of endometriosis and its control. Hum Reprod Update. 2009 Jul-Aug;15(4):441-61. doi: 10.1093/humupd/dmp007. Epub 2009 Mar 11. PMID 19279046
- [Background] Mabrouk M, Spagnolo E, Raimondo D, D'Errico A, Caprara G, Malvi D, Catena F, Ferrini G, Paradisi R, Seracchioli R. Segmental bowel resection for colorectal endometriosis: is there a correlation between histological pattern and clinical outcomes? Hum Reprod. 2012 May;27(5):1314-9. doi: 10.1093/humrep/des048. Epub 2012 Mar 12. PMID 22416007
- See also: Related Info — http://www.dexeus.com